CLINICAL TRIAL: NCT00194779
Title: A Study of Weekly Doxorubicin and Daily Oral Cyclophosphamide Plus G-CSF Followed by Weekly Paclitaxel as Neoadjuvant Therapy for Resectable, Hormone Receptor Negative or Hormone Receptor Positive, HER-2/Neu Positive Breast Cancer Followed by a Novel Regimen of Capecitabine, Methotrexate and Vinorelbine for Patients Who Do Not Have Either a Macroscopic or Microscopic Pathologic Complete Response, a Phase II Study
Brief Title: Combination Chemotherapy and Filgrastim Before Surgery in Treating Patients With HER2-Positive Breast Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hannah Linden, Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6278; NCI-2011-00934 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Results first posted 2018-03-12 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Estrogen Receptor-negative Breast Cancer; Estrogen Receptor-positive Breast Cancer; HER2-positive Breast Cancer; Progesterone Receptor-negative Breast Cancer; Progesterone Receptor-positive Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel; Taxes; Filgrastim; Granulocyte Colony-Stimulating Factor; Capecitabine; Methotrexate; merphos; Vinorelbine; Biopsy, Needle; Immunohistochemistry; Trastuzumab; Tamoxifen; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (neoadjuvant therapy, adjuvant therapy) (Experimental): See Detailed Description.
  Interventions: Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Drug: paclitaxel; Biological: filgrastim; Drug: capecitabine; Drug: methotrexate; Drug: vinorelbine tartrate; Procedure: needle biopsy; Procedure: therapeutic conventional surgery; Other: immunohistochemistry staining method; Biological: trastuzumab; Drug: tamoxifen citrate; Drug: letrozole; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given PO
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Drug: capecitabine — Given PO
  Other Names: CAPE; Ro 09-1978/000; Xeloda
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: vinorelbine tartrate — Given IV
  Other Names: Eunades; navelbine ditartrate; NVB; VNB
Procedure: needle biopsy — Correlative studies
  Other Names: aspiration biopsy; puncture biopsy
Procedure: therapeutic conventional surgery — Undergo definitive breast surgery
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Drug: tamoxifen citrate — Given PO
  Other Names: Nolvadex; TAM; tamoxifen; TMX
Drug: letrozole — Given PO
  Other Names: CGS 20267; Femara; LTZ
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving combination chemotherapy and filgrastim together before surgery works in treating patients with human epidermal growth receptor 2 (HER2)-positive breast cancer that can be removed by surgery. Drugs used in chemotherapy, such as doxorubicin hydrochloride, cyclophosphamide, and paclitaxel work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving combination chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Colony-stimulating factors, such as filgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving doxorubicin hydrochloride, cyclophosphamide, and filgrastim together followed by paclitaxel before surgery may be an effective treatment for breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the pathologic response rate in patients with operable breast cancer treated with a two part, neoadjuvant regimen consisting of weekly doxorubicin (doxorubicin hydrochloride) and daily oral cyclophosphamide given with G-CSF (filgrastim) support for 12 weeks followed weekly paclitaxel for 12 weeks.

SECONDARY OBJECTIVES:

I. To assess the clinical response rate in patients with surgically resectable breast cancer treated with weekly doxorubicin and daily oral cyclophosphamide given with G-CSF support for 12 weeks.

II. To assess the clinical response rate in patients with surgically resectable breast cancer treated with weekly paclitaxel for 12 weeks.

III. To assess the relapse rate, overall and disease-free survival in patients with operable breast cancer treated with neoadjuvant chemotherapy consisting of weekly doxorubicin and daily oral cyclophosphamide given with G-CSF support for 12 weeks followed weekly paclitaxel for 12 weeks and adjuvant chemotherapy with Xeloda (capecitabine), Methotrexate and Navelbine (vinorelbine tartrate) (XMN).

IV. To assess the toxicity associated with these regimens. V. To assess whether the phenotype of breast cancer changes with treatment. VI. To assess whether phenotypic changes in breast tumors predict outcome.

OUTLINE:

PART I: Patients receive doxorubicin hydrochloride intravenously (IV) on day 1 of each week, cyclophosphamide orally (PO) once daily (QD), and filgrastim subcutaneously (SC) QD on days 2-7 of each week. Treatment continues for 12 weeks in the absence of disease progression or unacceptable toxicity.

PART II: Patients* receive paclitaxel IV over 1 hour on day 1 of each week. Treatment continues for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo definitive surgical resection by partial mastectomy (lumpectomy) or mastectomy after completion of neoadjuvant chemotherapy.

PART III: Patients** unable to achieve complete pathologic response (pCR) or disease that has been down-staged to =< 1 cm with no positive nodes following surgery receive capecitabine PO twice daily (BID) on days 1-14, methotrexate IV on days 1, 8 and 15, and vinorelbine tartrate IV over 6-10 minutes on days 1, 8, and 15. Treatment repeats every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients with HER2/neu-positive disease also receive trastuzumab IV over 30-90 minutes once weekly or every 3 weeks for 1 year beginning in Part II.

NOTE: **Patients with hormone receptor-positive disease also receive tamoxifen PO QD for 5 years (premenopausal) OR letozole PO QD or tamoxifen PO QD for 5 years (postmenopausal) beginning in Part III.

After completion of study treatment, patients are followed up every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Have known tumor HER-2/neu expression; if determination is "intermediate" by immunohistochemistry, fluorescent in situ hybridization (FISH) must be performed; protocol therapy is determined by HER-2/neu result
* Have histologically confirmed, operable breast cancer that is either:
* Hormone receptor (estrogen receptor [ER] or progesterone receptor [PR]) positive and HER2/neu positive or
* ER/PR negative
* Have radiographically measurable breast cancer > 1cm (Operable lesions are T1c-T3 and N0-N2a; histologic confirmation should be by core needle biopsy only)
* Be chemotherapy naïve
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Absolute neutrophil count (ANC) >= 1,500
* Platelet count >= 100,000
* Serum creatinine =< 1.5 x international upper limit of normal (IULN)
* Bilirubin < 2.0
* Serum glutamic oxaloacetic transaminase (SGOT)/serum glutamic pyruvate transaminase (SGPT) =< 2 x IULN
* Alkaline phosphatase =< 2 x IULN
* Have staging studies and tumor assessment prior to registration; staging studies include physical exam with bidimensional tumor measurements and mammography, ultrasound, or magnetic resonance imaging (MRI) to assess tumor volume; sentinel lymph node dissection or axillary needle biopsy must be completed prior to enrollment; MRI and positron emission tomography (PET) (fluorodeoxyglucose [FDG], methoxyisobutylisonitrile [MIBI] and fluoroestradiol [FES]) imaging will be done before enrollment if clinically indicated to assess tumor volume or may be done within the first month of study participation on another institutional protocol
* Patients with clinically apparent cardiac disease, or history of same, are not eligible; patients who are >= 60 years of age or who have a history of hypertension must have an echocardiogram or multi gated acquisition scan (MUGA) prior to enrollment; patients with breast cancer that is HER-2/neu positive who will receive herceptin (trastuzumab) must have an echocardiogram or MUGA scan; the left ventricular ejection fraction (LVEF) must be within the institutional normal range; if LVEF is > 75%, the investigator should consider having the LVEF reviewed or repeating the MUGA prior to registration
* Women of childbearing potential must have a negative pregnancy test within seven days prior to registration
* Be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study specific screening procedures

Exclusion Criteria:

* Primary tumor =< 1 cm, not measurable; inflammatory disease
* Pregnant or lactating; woman of childbearing potential with either a positive or no pregnancy test at baseline are excluded; postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential; patients must agree to continue contraception for 30 days from the date of the last study drug administration; woman of childbearing potential not using a reliable and appropriate contraceptive method are excluded
* Evidence of distant metastatic disease
* Prior chemotherapy or hormonal therapy for breast cancer
* Except for the following no other malignancy is allowed: synchronous ipsilateral breast cancer of the same subtype (ER/PR, HER-2/neu), adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer or other stage I or II cancer from which the patient has been disease free for at least 5 years
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known sensitivity to 5-fluorouracil
* Previous enrollment in an investigational drug study within the past four weeks
* History of uncontrolled seizures, central nervous system disorders, or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance with oral drug intake
* Patients with cardiac disease that would preclude the use of Adriamycin, Taxol or Herceptin are not eligible
* Active cardiac disease:
* Angina pectoris that requires the use of antianginal medication
* Cardiac arrhythmia requiring medication
* Severe conduction abnormality
* Clinically significant valvular disease
* Cardiomegaly on chest x-ray
* Ventricular hypertrophy on electrocardiogram (EKG)
* Uncontrolled hypertension, (diastolic greater than 100 mm/Hg or systolic > 200 mm/hg)
* Current use of digitalis or beta blockers for congestive heart failure (CHF)
* Clinically significant pericardial effusion
* History of cardiac disease:
* Myocardial infarction documented as a clinical diagnosis or by EKG or any other test
* Documented congestive heart failure
* Documented cardiomyopathy
* Documented arrhythmia or cardiac valvular disease that requires medication or is medically significant
* Major surgery within 4 weeks of the start of study treatment without complete recovery
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Known, existing uncontrolled coagulopathy
* Unwillingness to give written informed consent
* Unwillingness to participate or inability to comply with the protocol for the duration of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-10; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgiana Ellis, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] — Population: Age data is missing from 5 patients
  years
    number analyzed (Participants) | 45
    (all) | 47 [27 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 35
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Combined Rate of Microscopic pCR and Macroscopic Pathologic Complete Response (mCR)
Description: Microscopic pCR: No evidence of microscopic invasive tumor at the primary site or in the regional lymph nodes at the time of definitive surgical resection. mCR: The examining pathologist cannot identify gross residual tumor mass in the surgical specimen. This differs from a pCR where the specimen must also be negative for invasive tumor by microscopy. For this study, we are using a definition of mCR that will make the trial more translatable to other institutions. For this study, mCR will be defined as no focus of invasive cancer >= 1 cm.
  Count of participants with either a pCR or mCR.
Time Frame: Up to 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Number analyzed (Participants) | 42
Participants | 29

2. Secondary Outcome: Number and Percent of Patients Reporting Grade 2, 3, 4, or Fatal Toxicities of These Regimens, Need for Dose Reduction, or Treatment Interruption or Discontinuation
Time Frame: From the initiation of study treatments to 30 days after the end of neoadjuvant treatment or adjuvant treatment if received
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Number analyzed (Participants) | 46
Participants | 32

3. Secondary Outcome: Correlation of Molecular Markers With Response
Time Frame: After completion of neoadjuvant therapy
Population: Due to lack of funding, none of the tissue specimens from participants were tested for EGFR, AR, P53 and Topo2alpha expression, as originally intended by the protocol.
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Number analyzed (Participants) | 0

4. Secondary Outcome: Relapse Rate in Patients With Operable Breast Cancer Treated With Neoadjuvant Chemotherapy for 12 Weeks Followed by Weekly Paclitaxel for 12 Weeks and Adjuvant Chemotherapy
Description: Count of patients that relapsed.
Time Frame: Up to 8 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Number analyzed (Participants) | 31
Participants | 7

5. Secondary Outcome: Time to Progression
Description: Median time to progression free survival.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Number analyzed (Participants) | 31
months | NA [NA to NA] — Median progression-free survival time was not reached because there were too few events (relapses/deaths).

6. Secondary Outcome: OS in Patients With Operable Breast Cancer Treated With Neoadjuvant Chemotherapy for 12 Weeks Followed Weekly Paclitaxel for 12 Weeks and Adjuvant Chemotherapy With XMN
Description: Kaplan-Meier estimate of overall survival, assessed at 1, 2, and 5 years.
Time Frame: 1, 2, and 5 years
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Number analyzed (Participants) | 31
survival probability
  1 year | 1 [1 to 1]
  2 years | .94 [.85 to 1]
  5 years | .90 [.81 to 1]

7. Secondary Outcome: Disease-free Survival
Description: Kaplan-Meier estimate of disease-free survival, assessed at 1, 2, and 5 years.
Time Frame: 1, 2, and 5 years
Measure: Number (95% Confidence Interval); unit: disease-free survival probability
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Number analyzed (Participants) | 31
disease-free survival probability
  1 year | .97 [.91 to 1]
  2 years | .90 [.81 to 1]
  5 years | .84 [.72 to .98]

8. Secondary Outcome: Clinical Response to Neoadjuvant Therapy
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Number analyzed (Participants) | 47
Participants
  CR | 6
  PR | 33
  SD | 6
  ND | 2

9. Secondary Outcome: Clinical Response to Paclitaxel
Time Frame: Up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Number analyzed (Participants) | 45
Participants
  CR | 23
  PR | 14
  SD | 4
  ND | 3
  Progression | 1

ADVERSE EVENTS:
Arm/Group | Treatment (Neoadjuvant Therapy, Adjuvant Therapy)
Serious Adverse Events (participants affected / at risk) | 8/50
Other Adverse Events (participants affected / at risk) | 40/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Neoadjuvant Therapy, Adjuvant Therapy) (N=50)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Depression (Psychiatric disorders) | 1
Neutropenia (Investigations) | 5
Death (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Neoadjuvant Therapy, Adjuvant Therapy) (N=50)
Leukocytes Decreased (Blood and lymphatic system disorders) | 32
Neutropenic Fever (Blood and lymphatic system disorders) | 4
Numbness (lymphs) (Blood and lymphatic system disorders) | 32
Pain (lymphs) (Blood and lymphatic system disorders) | 29
Pain (chest) (Cardiac disorders) | 12
Palpitations (Cardiac disorders) | 29
Tachycardia (Cardiac disorders) | 11
Clear Drainage (ear) (Ear and labyrinth disorders) | 20
Blurred Vision (Eye disorders) | 19
Dry Eyes (Eye disorders) | 26
Swollen Eyes (Eye disorders) | 16
Watery Eyes (Eye disorders) | 7
Constipation (Gastrointestinal disorders) | 28
Cramping (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 12
Dry Mouth (Gastrointestinal disorders) | 20
Dysgeusia (Gastrointestinal disorders) | 15
Dysphagia (Gastrointestinal disorders) | 10
Esophagitis (Gastrointestinal disorders) | 14
Flatulence (Gastrointestinal disorders) | 9
Bleeding gums (while brushing) (Gastrointestinal disorders) | 4
Heartburn (Gastrointestinal disorders) | 12
Irritable Bowel Syndrome (Gastrointestinal disorders) | 6
Metallic taste (Gastrointestinal disorders) | 10
Mucositis (oral/stomatitis) (Gastrointestinal disorders) | 31
Nausea (Gastrointestinal disorders) | 9
Oral Herpes (Gastrointestinal disorders) | 4
Pain (teeth) (Gastrointestinal disorders) | 3
Reflux (Gastrointestinal disorders) | 5
Stomach Flu (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 7
Alopecia (General disorders) | 7
Fatigue (General disorders) | 12
Hot flashes (General disorders) | 3
Pain (General disorders) | 3
Pain (bone) (General disorders) | 5
Swelling (joints) (General disorders) | 4
Weight loss (General disorders) | 4
Acute infusion allergic reaction (Immune system disorders) | 3
Urinary tract infection (Infections and infestations) | 4
Hemoglobin decreased (Investigations) | 3
Ion gap decreased (Investigations) | 29
Lactate dehydrogenase increased (Investigations) | 36
Lymphopenia Decreased (Investigations) | 8
Neutrophils Decreased (Investigations) | 30
Platelets decreased (Investigations) | 27
Platelets increased (Investigations) | 11
SGOT increased (Investigations) | 11
SGPT increased (Investigations) | 5
Urea nitrogen decreased (Investigations) | 19
Weight gain (Investigations) | 24
Anorexia (Metabolism and nutrition disorders) | 5
Calcium decreased (Metabolism and nutrition disorders) | 4
Ferritin increased (Metabolism and nutrition disorders) | 14
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 14
Athralgia (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness (Musculoskeletal and connective tissue disorders) | 15
Pain (joint) (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 15
Paresthesia (Nervous system disorders) | 3
Vertigo (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 9
Chemo brain (Psychiatric disorders) | 5
Confusion (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 9
Memory loss (Psychiatric disorders) | 4
Incontinence (urinary) (Renal and urinary disorders) | 3
Vaginal discharge (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3
Dry sweats (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3
Hand foot syndrome (Skin and subcutaneous tissue disorders) | 8
Hyperpigmintation (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 3
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes